CLINICAL TRIAL: NCT00984711
Title: A Phase IV, Post-marketing, Observational Study of Rituxan in Rheumatoid Arthritis Patients in Routine Clinical Practice
Brief Title: Observational Study of Rituxan in Rheumatoid Arthritis Patients in Routine Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PerCuro Clinical Research Ltd (Other)
Responsible Party: Christopher Atkins MD, PerCuro Clinical Research Ltd.
Other Study IDs: ML21427
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was designed to gather data regarding the efficacy and safety of Rituxan in clinical practice whereby patients may present with concomitant medical conditions, medications as well as varying presentations of rheumatoid arthritis not always captured within the "purer" population seen in an industry sponsored clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active rheumatoid arthritis as defined by ACR criteria
* > 18 years of age at time of consent
* Able to start RITUXAN therapy per the approved product monograph within approximately 30 days of confirmed enrollment

Exclusion Criteria:

* Known Type 1 hypersensitivity or anaphylactic reactions to murine proteins, Chinese Hamster Ovary cell proteins or to any component of RITXAN as per approved Product monograph
* Presence of any significant and or uncontrolled medical condition, which in the Investigator's opinion, precludes the use of RITUXAN as outlined in the Product Monograph

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with active rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Atkins, MD, Principal Investigator — PerCuro Clinical Research Ltd
Locations (1):
- PerCuro Clinical Research Ltd., Victoria, British Columbia, Canada